CLINICAL TRIAL: NCT03551496
Title: A Randomized Trial Comparing the Drug-Eluting Stent (DES) Below-the-Knee (BTK) Vascular Stent System (DES BTK Vascular Stent System) vs Percutaneous Transluminal Angioplasty (PTA) Treating Infrapopliteal Lesions in Subjects With Critical Limb Ischemia
Brief Title: The DES BTK Vascular Stent System vs PTA in Subjects With Critical Limb Ischemia
Acronym: SAVAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S2348
Record Dates: First submitted 2018-05-15; First posted 2018-06-11 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Intervention Model Description: Approximately 201 subjects will be randomized in a 2:1 fashion for phase A RCT. Randomizations will be stratified by investigational center and lesion length with 2 subjects receiving the DES BTK for every 1 subject receiving treatment with standard PTA.
Who Masked: Outcomes Assessor
Masking Description: A review of the wound assessment data will be completed by independent reviewer(s) who will be blinded to the randomized therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- DES BTK (Experimental): Treatment with DES BTK
  Interventions: Combination Product: Drug Eluting Stent - Below the Knee
- Conventional PTA (Active Comparator): Treatment with standard PTA
  Interventions: Device: Standard PTA Control Arm

INTERVENTIONS:
Combination Product: Drug Eluting Stent - Below the Knee — Treatment arm with DES-BTK, starting with one size of the device - 3.5 mm X 80 mm
  Arms: DES BTK
Device: Standard PTA Control Arm — The PTA device used must be market-released in the investigational center's geography and the size (ie, diameter, balloon length and catheter length) will be determined by the investigator.
  Arms: Conventional PTA

SUMMARY:
Single phased global, prospective, multicenter clinical trial designed to demonstrate a superior patency rate and acceptable safety in below the knee arteries with lesions treated with the DES BTK Vascular Stent System vs. percutaneous transluminal angioplasty (PTA).

DETAILED DESCRIPTION:
A global, prospective, multicenter, 2:1 randomized trial evaluating the safety and effectiveness of the DES BTK Vascular Stent System compared to standard percutaneous transluminal angioplasty to treat infrapopliteal artery lesions in subjects with critical limb ischemia(CLI).

Approximately 201 subjects will be randomized/enrolled to support a 2:1 randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years or older and has signed and dated the trial informed consent form (ICF)
2. Subject is willing and able to comply with the trial testing, procedures and follow-up schedule
3. Subject has chronic, symptomatic lower limb ischemia, determined by Rutherford categories 4 or 5 in the target limb, with wound(s) confined to toes/forefoot
4. Subject is a male or non-pregnant female. If female of child-bearing potential, and if sexually active must be using, or agree to use, a medically-acceptable method of birth control as confirmed by the investigator

Intra-procedure Inclusion Criteria:

1. Stenotic, restenotic or occlusive target lesion(s) located in the tibioperoneal trunk, anterior tibial, posterior tibial and/or peroneal artery(ies).
2. Target lesion(s) must be at least 4cm above the ankle joint
3. A single target lesion per vessel, in up to 2 vessels, in a single limb
4. Degree of stenosis ≥ 70% by visual angiographic assessment
5. Reference vessel diameter is between 2.5 - 3.25mm for phase A RCT
6. Total target lesion length (or series of lesion segments) to be treated is ≤ 70 mm for phase A RCT prior to the data monitoring committee's approval for stent overlap. (Note: Lesion segment(s) must be fully covered with one DES BTK stent, if randomized to stent)
7. Total target lesion length (or series of lesion segments) to be treated is ≤ 140 mm for phase A RCT after the data monitoring committee's approval for stent overlap (Note: Lesion segment(s) must be fully covered with up to two DES BTK stents, if randomized to stent)
8. Target vessel(s) reconstitute(s) at or above the stenting limit zone (4cm above the ankle joint)
9. Target lesion(s) is located in an area that may be stented without blocking access to patent main branches
10. Treatment of all above the knee inflow lesion(s) is successful prior to treatment of the target lesion
11. Guidewire has successfully crossed the target lesion(s)

Exclusion Criteria:

1. Life expectancy ≤ 1year
2. Stroke ≤ 90 days prior to the procedure date
3. Prior or planned major amputation in the target limb
4. Previous surgery in the target vessel(s) (including prior ipsilateral crural bypass)
5. Previously implanted stent in the target vessel(s)
6. Failed PTA of target lesion/vessel ≤ 60 days prior to the procedure date
7. Renal failure as measured by a GFR ≤ 30ml/min per 1.73m2, measured ≤ 30 days prior to the procedure date
8. Subject has a platelet count ≤ 50 or ≥ 600 X 103/µL ≤ 30 days prior to the procedure date
9. NYHA class IV heart failure
10. Subject has symptomatic coronary artery disease (ie, unstable angina)
11. History of myocardial infarction or thrombolysis ≤ 90 days prior to the procedure date
12. Non-atherosclerotic disease resulting in occlusion (eg, embolism, Buerger's disease, vasculitis)
13. Subject is currently taking Canagliflozin
14. Body Mass Index (BMI) <18
15. Active septicemia or bacteremia
16. Coagulation disorder, including hypercoagulability
17. Contraindication to anticoagulation or antiplatelet therapy
18. Known allergies to stent or stent components
19. Known allergy to contrast media that cannot be adequately pre-medicated prior to the interventional procedure
20. Known hypersensitivity to heparin
21. Subject is on a high dose of steroids or is on immunosuppressive therapy
22. Subject is currently participating, or plans to participate in, another investigational trial that may confound the results of this trial (unless written approval is received from the Boston Scientific study team)

Intra-procedure Exclusion Criteria

1. Angiographic evidence of intra-arterial acute/subacute thrombus or presence of atheroembolism
2. Treatment required in > 2 target vessels (Note: a target lesion originating in one vessel and extending into another vessel is considered 1 target vessel)
3. Treatment requires the use of alternate therapy in the target vessel(s)/lesion(s), (eg, atherectomy, cutting balloon, re-entry devices, laser, radiation therapy)
4. Aneurysm is present in the target vessel(s)
5. Extremely calcified lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2023-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jihad Mustapha, MD, Principal Investigator — Advanced Cardiac & Vascular Centers for Amputation Prevention; Hendrik van Overhagen, MD, Principal Investigator — HAGA Ziekenhuis (HagaZiekenhuis van Den Haag); Patrick Geraghty, MD, Principal Investigator — Washington University School of Medicine; Masato Nakamura, MD, PhD, Principal Investigator — Toho University Ohashi Medical Center - Division of Cardiovascular Medicine
Locations (42):
- United States (26):
  - St. Bernards Medical Center, Jonesboro, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - University of California, San Francisco, San Francisco, California
  - Colorado VA, Denver, Colorado
  - Bradenton Cardiology, Bradenton, Florida
  - Willis Knighton Bossier Medical Center - Grace Research, LLC, Bossier City, Louisiana
  - Cardiovascular Institute of the South Clinical Research Corporation, Houma, Louisiana
  - Advanced Cardiac & Vascular Centers for Amputation Prevention, Grand Rapids, Michigan
  - United Heart and Vascular Clinic, Saint Paul, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - New Mexico Heart Institute, PA, Albuquerque, New Mexico
  - New York University Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Amputation Prevention Center of North Carolina, Cary, North Carolina
  - NC Heart and Vascular Research, LLC, Raleigh, North Carolina
  - Wake Medical Center, Raleigh, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - OhioHealth Research and Innovation Institute - Riverside Methodist Hospital, Columbus, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Saint Vincent Consultants in Cardiovascular Diseases at St. Vincent Hospital, Erie, Pennsylvania
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Heart Hospital of Austin, Austin, Texas
  - Texas Tech University Health, Lubbock, Texas
  - THR Presbyterian Plano, Plano, Texas
- Belgium (3):
  - AZ Sint-Blasius, Dendermonde
  - ZOL Genk (Ziekenhuis Oost-Limburg), Genk
  - UZ Gent (Universitair Ziekenhuis Gent), Ghent
- France (4):
  - CHU Nantes, Nantes
  - Hopital Paris Saint Joseph, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Clinique Pasteur, Toulouse
- Japan (8):
  - Tokyo Bay Urayasu Ichikawa Medical Center, Urayasu-shi, Chiba
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Asahikawa Medical University Hospital, Asahikawa-shi, Hokkaido
  - Kansai Rosai Hospital, Amagasaki, Hyōgo
  - Nara Medical University Hospital, Kashihara, Nara
  - Kishiwada Tokushukai Hospital, Kishiwada, Osaka
  - Tokyo Medical and Dental University, Medical Hospital, Bunkyō-Ku, Tokyo
  - Toho University Ohashi Medical Center, Meguro City, Tokyo
- HAGA Ziekenhuis (Haga Ziekenhuis van Den Haag), The Hague, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kolte D, Kennedy KF, Shishehbor MH, Abbott JD, Khera S, Soukas P, Mamdani ST, Hyder ON, Drachman DE, Aronow HD. Thirty-Day Readmissions After Endovascular or Surgical Therapy for Critical Limb Ischemia: Analysis of the 2013 to 2014 Nationwide Readmissions Databases. Circulation. 2017 Jul 11;136(2):167-176. doi: 10.1161/CIRCULATIONAHA.117.027625. Epub 2017 May 2. PMID 28465288
- [Background] Conte MS, Geraghty PJ, Bradbury AW, Hevelone ND, Lipsitz SR, Moneta GL, Nehler MR, Powell RJ, Sidawy AN. Suggested objective performance goals and clinical trial design for evaluating catheter-based treatment of critical limb ischemia. J Vasc Surg. 2009 Dec;50(6):1462-73.e1-3. doi: 10.1016/j.jvs.2009.09.044. Epub 2009 Nov 7. PMID 19897335
- [Background] Scheinert D, Katsanos K, Zeller T, Koppensteiner R, Commeau P, Bosiers M, Krankenberg H, Baumgartner I, Siablis D, Lammer J, Van Ransbeeck M, Qureshi AC, Stoll HP; ACHILLES Investigators. A prospective randomized multicenter comparison of balloon angioplasty and infrapopliteal stenting with the sirolimus-eluting stent in patients with ischemic peripheral arterial disease: 1-year results from the ACHILLES trial. J Am Coll Cardiol. 2012 Dec 4;60(22):2290-5. doi: 10.1016/j.jacc.2012.08.989. PMID 23194941
- [Background] Spreen MI, Martens JM, Hansen BE, Knippenberg B, Verhey E, van Dijk LC, de Vries JP, Vos JA, de Borst GJ, Vonken EJ, Wever JJ, Statius van Eps RG, Mali WP, van Overhagen H. Percutaneous Transluminal Angioplasty and Drug-Eluting Stents for Infrapopliteal Lesions in Critical Limb Ischemia (PADI) Trial. Circ Cardiovasc Interv. 2016 Feb;9(2):e002376. doi: 10.1161/CIRCINTERVENTIONS.114.002376. PMID 26861113
- [Background] Kinlay S. Management of Critical Limb Ischemia. Circ Cardiovasc Interv. 2016 Feb;9(2):e001946. doi: 10.1161/CIRCINTERVENTIONS.115.001946. PMID 26858079
- [Background] Elsayed S, Clavijo LC. Critical limb ischemia. Cardiol Clin. 2015 Feb;33(1):37-47. doi: 10.1016/j.ccl.2014.09.008. PMID 25439329
- [Background] Conte MS. Critical appraisal of surgical revascularization for critical limb ischemia. J Vasc Surg. 2013 Feb;57(2 Suppl):8S-13S. doi: 10.1016/j.jvs.2012.05.114. PMID 23336860
- [Background] Gray BH, Diaz-Sandoval LJ, Dieter RS, Jaff MR, White CJ; Peripheral Vascular Disease Committee for the Society for Cardiovascular Angiography and Interventions. SCAI expert consensus statement for infrapopliteal arterial intervention appropriate use. Catheter Cardiovasc Interv. 2014 Oct 1;84(4):539-45. doi: 10.1002/ccd.25395. Epub 2014 Jul 18. PMID 25045160
- [Background] Adam DJ, Beard JD, Cleveland T, Bell J, Bradbury AW, Forbes JF, Fowkes FG, Gillepsie I, Ruckley CV, Raab G, Storkey H; BASIL trial participants. Bypass versus angioplasty in severe ischaemia of the leg (BASIL): multicentre, randomised controlled trial. Lancet. 2005 Dec 3;366(9501):1925-34. doi: 10.1016/S0140-6736(05)67704-5. PMID 16325694
- [Background] Popplewell MA, Davies HOB, Narayanswami J, Renton M, Sharp A, Bate G, Patel S, Deeks J, Bradbury AW. A Comparison of Outcomes in Patients with Infrapopliteal Disease Randomised to Vein Bypass or Plain Balloon Angioplasty in the Bypass vs. Angioplasty in Severe Ischaemia of the Leg (BASIL) Trial. Eur J Vasc Endovasc Surg. 2017 Aug;54(2):195-201. doi: 10.1016/j.ejvs.2017.04.020. Epub 2017 Jun 8. PMID 28602580
- [Background] Sadaghianloo N, Jean-Baptiste E, Declemy S, Mousnier A, Brizzi S, Hassen-Khodja R. Percutaneous angioplasty of long tibial occlusions in critical limb ischemia. Ann Vasc Surg. 2013 Oct;27(7):894-903. doi: 10.1016/j.avsg.2013.02.008. PMID 23993107
- [Background] Bosiers M, Scheinert D, Peeters P, Torsello G, Zeller T, Deloose K, Schmidt A, Tessarek J, Vinck E, Schwartz LB. Randomized comparison of everolimus-eluting versus bare-metal stents in patients with critical limb ischemia and infrapopliteal arterial occlusive disease. J Vasc Surg. 2012 Feb;55(2):390-8. doi: 10.1016/j.jvs.2011.07.099. Epub 2011 Dec 14. PMID 22169682
- [Background] Spreen MI, Martens JM, Knippenberg B, van Dijk LC, de Vries JPM, Vos JA, de Borst GJ, Vonken EPA, Bijlstra OD, Wever JJ, Statius van Eps RG, Mali WPTM, van Overhagen H. Long-Term Follow-up of the PADI Trial: Percutaneous Transluminal Angioplasty Versus Drug-Eluting Stents for Infrapopliteal Lesions in Critical Limb Ischemia. J Am Heart Assoc. 2017 Apr 14;6(4):e004877. doi: 10.1161/JAHA.116.004877. PMID 28411244
- [Background] de Weger VA, Beijnen JH, Schellens JH. Cellular and clinical pharmacology of the taxanes docetaxel and paclitaxel--a review. Anticancer Drugs. 2014 May;25(5):488-94. doi: 10.1097/CAD.0000000000000093. PMID 24637579
- [Background] Ng VG, Mena C, Pietras C, Lansky AJ. Local delivery of paclitaxel in the treatment of peripheral arterial disease. Eur J Clin Invest. 2015 Mar;45(3):333-45. doi: 10.1111/eci.12407. Epub 2015 Feb 14. PMID 25615282
- [Background] Dake MD, Van Alstine WG, Zhou Q, Ragheb AO. Polymer-free paclitaxel-coated Zilver PTX Stents--evaluation of pharmacokinetics and comparative safety in porcine arteries. J Vasc Interv Radiol. 2011 May;22(5):603-10. doi: 10.1016/j.jvir.2010.12.027. Epub 2011 Mar 17. PMID 21419649
- [Background] Banerjee S, Sarode K, Mohammad A, Gigliotti O, Baig MS, Tsai S, Shammas NW, Prasad A, Abu-Fadel M, Klein A, Armstrong EJ, Jeon-Slaughter H, Brilakis ES, Bhatt DL. Femoropopliteal Artery Stent Thrombosis: Report From the Excellence in Peripheral Artery Disease Registry. Circ Cardiovasc Interv. 2016 Feb;9(2):e002730. doi: 10.1161/CIRCINTERVENTIONS.115.002730. PMID 26839391
- [Background] Federman DG, Ladiiznski B, Dardik A, Kelly M, Shapshak D, Ueno CM, Mostow EN, Richmond NA, Hopf HW. Wound Healing Society 2014 update on guidelines for arterial ulcers. Wound Repair Regen. 2016 Jan-Feb;24(1):127-35. doi: 10.1111/wrr.12395. No abstract available. PMID 26663663
- [Derived] van Overhagen H, Nakamura M, Geraghty PJ, Rao S, Arroyo M, Soga Y, Iida O, Armstrong E, Nakama T, Fujihara M, Ansari MM, Mathews SJ, Goueffic Y, Jaff MR, Weinberg I, Pinto DS, Ohura N, Couch K, Mustapha JA. Primary results of the SAVAL randomized trial of a paclitaxel-eluting nitinol stent versus percutaneous transluminal angioplasty in infrapopliteal arteries. Vasc Med. 2023 Dec;28(6):571-580. doi: 10.1177/1358863X231199489. Epub 2023 Oct 16. PMID 37844137

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 201 enrolled participants, 201 met inclusion criteria and were randomized. Phase 2 was not conducted.
Period: Overall Study
Arm/Group | DES BTK | Conventional PTA
Started | 130 | 71
Completed | 114 | 61
Not Completed | 16 | 10
Not completed — Death | 11 | 7
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Other Reasons | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DES BTK | Conventional PTA | Total
Number analyzed (Participants) | 130 | 71 | 201
Age, Customized [Mean (Standard Deviation); unit: Years]
  Age (Year) | 73.27 (9.61) | 72.58 (10.14) | 73.02 (9.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 16 | 51
  Male | 95 | 55 | 150
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Hispanic or Latino | 7 | 4 | 11
  Race/Ethnicity: Caucasian | 69 | 35 | 104
  Race/Ethnicity: Asian | 33 | 18 | 51
  Race/Ethnicity: Black, of African heritage | 15 | 10 | 25
  Race/Ethnicity: Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  Race/Ethnicity: American Indian or Alaska Native | 1 | 1 | 2
  Race/Ethnicity: Other | 2 | 1 | 3
  Race/Ethnicity: Not Disclosed | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 80 | 45 | 125
  Japan | 33 | 17 | 50
  Europe | 17 | 9 | 26
Smoking [Count of Participants; unit: Participants]
  Current | 27 | 18 | 45
  Never | 36 | 18 | 54
  Previous | 66 | 35 | 101
  Unknown | 1 | 0 | 1
Current Diabetes Mellitus [Count of Participants; unit: Participants] | 87 | 47 | 134
History of Hyperlipidemia requiring medication [Count of Participants; unit: Participants] | 101 | 52 | 153
History of Hypertension requiring medication [Count of Participants; unit: Participants] | 115 | 59 | 174
History of Chronic Obstructive Pulmonary Disease [Count of Participants; unit: Participants] | 20 | 9 | 29
Cardiac History [Count of Participants; unit: Participants]
  History of Coronary Artery Disease | 75 | 40 | 115
  History of Myocardial Infarction (MI) | 29 | 13 | 42
  History of Congestive Heart Failure | 30 | 15 | 45
History of Percutaneous Coronary Intervention (PCI) [Count of Participants; unit: Participants] | 44 | 22 | 66
History of Coronary Artery Bypass Graft (CABG) Surgery [Count of Participants; unit: Participants] | 31 | 14 | 45
Current Anginal Status [Count of Participants; unit: Participants]
  Stable Angina | 22 | 9 | 31
  Unstable Angina | 0 | 0 | 0
  None | 108 | 62 | 170
  Unknown | 0 | 0 | 0
Neurologic/Renal History [Count of Participants; unit: Participants]
  History of Transient Ischemic Attacks (TIA) | 8 | 3 | 11
  History of Cerebrovascular Accident (CVA) | 17 | 11 | 28
  History of Renal Insufficiency | 23 | 11 | 34
  History of Renal Percutaneous Intervention | 3 | 0 | 3
History of amputation [Count of Participants; unit: Participants] | 28 | 16 | 44
History of amputation - Limb treated [Count of Participants; unit: Participants] — Population: 201 subjects analyzed; 44/201 subjects have a history of amputation
  Participants
    Target Limb: number analyzed (Participants) | 28 | 16 | 44
    Target Limb | 10 | 4 | 14
    Non-Target Limb: number analyzed (Participants) | 28 | 16 | 44
    Non-Target Limb | 16 | 9 | 25
    Both: number analyzed (Participants) | 28 | 16 | 44
    Both | 2 | 3 | 5
History of amputation - Type of amputation [Count of Participants; unit: Participants] — Population: 44/201 subjects have a history of amputation
  Participants
    Minor: number analyzed (Participants) | 28 | 16 | 44
    Minor | 23 | 13 | 36
    Major: number analyzed (Participants) | 28 | 16 | 44
    Major | 6 | 4 | 10
History of other peripheral vascular surgery [Count of Participants; unit: Participants] | 14 | 11 | 25
History of other peripheral vascular surgery - Limb Treated [Count of Participants; unit: Participants] — Population: 25/201 subjects have a history of other peripheral vascular surgery
  Participants
    Target Limb: number analyzed (Participants) | 14 | 11 | 25
    Target Limb | 4 | 4 | 8
    Non-Target Limb: number analyzed (Participants) | 14 | 11 | 25
    Non-Target Limb | 9 | 7 | 16
    Both: number analyzed (Participants) | 14 | 11 | 25
    Both | 1 | 0 | 1
History of other peripheral endovascular interventions with non-paclitaxel containing devices [Count of Participants; unit: Participants] | 82 | 37 | 119
History of other peripheral endovascular interventions with non-paclitaxel devices - Limb treated [Count of Participants; unit: Participants] — Population: 201 subjects analyzed; 119/201 subjects have a history of other peripheral endovascular interventions with non-paclitaxel containing devices
  Participants
    number analyzed (Participants) | 82 | 37 | 119
    Target Limb | 37 | 11 | 48
    Non-Target Limb | 27 | 18 | 45
    Both | 18 | 8 | 26
History of other peripheral endovascular with non-paclitaxel device-Type of most recent intervention [Count of Participants; unit: Participants] — Population: 119/201 subjects have a history of other peripheral endovascular interventions with non-paclitaxel containing devices. Multiple subjects had various interventions.
  Participants
    Atherectomy: number analyzed (Participants) | 82 | 37 | 119
    Atherectomy | 37 | 15 | 52
    Percutaneous Transluminal Angioplasty (PTA): number analyzed (Participants) | 82 | 37 | 119
    Percutaneous Transluminal Angioplasty (PTA) | 66 | 27 | 93
    Stenting: number analyzed (Participants) | 82 | 37 | 119
    Stenting | 35 | 15 | 50
    Other: number analyzed (Participants) | 82 | 37 | 119
    Other | 3 | 3 | 6
History of interventions with paclitaxel-containing devices [Count of Participants; unit: Participants] | 59 | 29 | 88

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Primary Patency
Description: Twelve-Month Primary Patency defined as a binary endpoint to be determined via duplex ultrasound (DUS) measuring flow at the 12-month follow-up visit, in the absence of clinically-driven target lesion revascularization (TLR) or bypass of the target lesion. Data table consists of the number of participants with flow as assessed by DUS.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | DES BTK | Conventional PTA
Number analyzed (Participants) | 103 | 50
Participants | 70 | 38

2. Primary Outcome: Number of Participants Free From Major Adverse Events (MAE)
Description: The primary safety endpoint assesses freedom from major adverse events (MAE) at 12 months post-procedure. (MAE is defined as: above ankle amputation in index limb; major re-intervention; and perioperative (30 day) mortality)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | DES BTK | Conventional PTA
Number analyzed (Participants) | 119 | 64
Participants | 109 | 61

3. Other Pre Specified Outcome: Number of Participants With Assisted Primary Patency
Description: Assisted primary patency defined as the percentage (%) of lesions without clinically-driven TLR and those with clinically-driven TLR (not due to complete occlusion or by-pass) which show flow by DUS without restenosis.
Time Frame: 12 months post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | DES BTK | Conventional PTA
Number analyzed (Participants) | 91 | 44
Participants | 75 | 41

4. Other Pre Specified Outcome: Number of Participants With Clinically Driven Target Lesion Revascularization
Description: Clinically-driven target lesion revascularization is defined as any surgical or percutaneous intervention to the target lesion after the index procedure if:
  1. Occurring within 5mm proximal or distal to the original treatment segment with diameter stenosis ≥50% by quantitative angiography and if participant has recurrent symptoms OR
  2. In-lesion diameter stenosis less than 50% might also be considered a MAE by the CEC if the subject has recurrent symptoms.
  Recurrent symptoms are defined as having ≥ 1 change in Rutherford Classification or associated with decreased ABI/TBI of ≥20% or ≥ 0.15 in the treated segment.
Time Frame: 12 months post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | DES BTK | Conventional PTA
Number analyzed (Participants) | 128 | 67
Participants | 21 | 10

5. Other Pre Specified Outcome: Number of Participants With Major Amputation (Defined as Amputation of the Lower Limb at the Ankle Level or Above)
Description: Rates of amputation of the lower limb at the ankle level or above
Time Frame: 12 months post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | DES BTK | Conventional PTA
Number analyzed (Participants) | 118 | 62
Participants | 3 | 1

6. Other Pre Specified Outcome: Participant Quality-of-Life Changes Via EuroQol 5 Dimension (EQ-5D) Questionnaire.
Description: The EQ-5D is a descriptive system of health-related quality-of-life states consisting of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take 1 of 5 responses. The responses record 5 levels of severity (no problems/slight problems/moderate problems/severe problems/extreme problems) within a particular EQ-5D dimension). The levels are assigned a numeric code 1-5 (eg, 1= no problems and 5= extreme problems).
Time Frame: 12 months post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | DES BTK | Conventional PTA
Number analyzed (Participants) | 99 | 53
Participants
  Mobility Improvement | 40 | 16
  Self-Care Improvement | 19 | 8
  Usual Activities Improvement | 32 | 17
  Pain/Discomfort Improvement | 48 | 18
  Anxiety/Depression Improvement | 28 | 12

7. Other Pre Specified Outcome: Participant Quality-of-Life Changes Via Vascular Quality of Life (VascuQol) Questionnaire.
Description: Changes in quality of life is measured using the Vascular Quality of Life (VascuQol) questionnaire, which is a 25 item questionnaire used to measure the quality-of-life in patients with lower limb ischemia. The tool is sub-divided into 5 domains: pain, symptoms, activities, social and emotional.
Time Frame: 12 months post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | DES BTK | Conventional PTA
Number analyzed (Participants) | 99 | 52
Participants
  Improvement in pain in leg (or foot) when walking | 61 | 27
  Improvement in worried that I might injure my leg | 42 | 21
  Improvement in cold feet have given | 50 | 26
  Improvement in ability to exercise or to play sports | 56 | 21
  Improvement in legs felt tired or weak | 55 | 26
  Improvement in restricted in spending time with friends or relatives | 44 | 18
  Improvement in pain in the foot (or leg) after going to bed at night | 58 | 31
  Improvement in pins and needles or numbness in leg (or foot) have caused | 53 | 26
  Improvement in the distance I can walk has improved | 39 | 17
  Improvement in ability to walk | 59 | 25
  Improvement in being (or becoming) housebound has concerned | 42 | 28
  Improvement in concerned about having poor circulation in legs | 68 | 26
  Improvement in pain in the foot (or leg) when resting | 67 | 31
  Improvement in ability to climb stairs | 47 | 20
  Improvement in ability to participate in social activities | 49 | 23
  Improvement in ability to do routine household work | 54 | 22
  Improvement in ulcers or sores on my leg (or foot) caused pain or distress | 45 | 15
  Improvement in the range of activities that would have liked to do | 58 | 26
  Improvement in problems caused by poor circulation made feel frustrated | 60 | 29
  Improvement in pain in the leg (or foot) given | 63 | 30
  Improvement in felt guilty about relying on friends or relatives | 47 | 28
  Improvement in ability to go shopping or carry bags | 50 | 21
  Improvement in worried in danger of losing a part of leg or foot | 58 | 28
  Improvement in distance I can walk became less | 48 | 25
  Improvement in depressed about the poor circulation in legs | 57 | 28

8. Other Pre Specified Outcome: Number of Participants With Baseline Wounds Assessed as Healed
Description: Wounds assessed for healed status by Independent Wound Assessors, blinded to randomized treatment.
Time Frame: 12 months post procedure
Population: Data for baseline wounds assessed as healed are based on subjects with the data point collected.
Measure: Count of Participants; unit: Participants
Arm/Group | DES BTK | Conventional PTA
Number analyzed (Participants) | 79 | 32
Participants | 34 | 15

9. Other Pre Specified Outcome: Number of Participants With Rate of Primary Sustained Clinical Improvement as Assessed by Changes in Rutherford Classification From Baseline
Description: Endpoint determined to be a success when there is an improvement in Rutherford Classification of one or more categories as compared to pre-procedure without the need for repeat TLR. Rutherford Classifications:
  i. Category 0 - Asymptomatic ii. Category 1 - Mild claudication iii. Category 2 - Moderate claudication iv. Category 3 - Severe claudication v. Category 4 - Ischemic rest pain vi. Category 5 - Minor tissue loss - nonhealing ulcer, focal gangrene vii. Category 6 - Major tissue loss - extending above transmetatarsal (TM) level
Time Frame: 12 months post procedure
Population: Data for Rate of Primary Sustained clinical Improvement as Assessed by Changes in Rutherford Classification from baseline are based on subjects with the data point collected
Measure: Count of Participants; unit: Participants
Arm/Group | DES BTK | Conventional PTA
Number analyzed (Participants) | 102 | 49
Participants | 80 | 36

10. Other Pre Specified Outcome: Number of Participants With Major, Serious, Non-serious, Unanticipated, Device-related and Procedure-related Adverse Events
Description: Adverse events (AEs) to be classified as major (defined as above ankle amputation of the index limb, major re-intervention (new bypass graft, jump/interposition graft, or thrombectomy/thrombolysis) and perioperative (30 day) mortality), serious, non-serious, unanticipated, procedure-related and device-related.
Time Frame: 12 months post procedure
Population: The data presented in this table for the serious, non-serious, unanticipated, device-related, and procedure-related events are based on crude event rates, and the data used for the major events is based on the subjects evaluable for the primary safety endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | DES BTK | Conventional PTA
Number analyzed (Participants) | 130 | 71
Participants
  Serious | 82 | 51
  Non serious | 84 | 37
  Major | 10 | 3
  Unanticipated | 0 | 0
  Device-Related | 16 | 6
  Procedure-Related | 21 | 16

11. Other Pre Specified Outcome: Number of Participants Who Were Admitted to the Hospital Within 30 Days After the Index Procedure.
Description: Hospitalizations related to Critical Limb Ischemia (CLI) due to target lesion revascularization (TLR)/target vessel revascularization (TVR) or Target Limb Major Amputation or Procedure/Device related Adverse Events
Time Frame: Up to 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | DES BTK | Conventional PTA
Number analyzed (Participants) | 130 | 71
Participants | 2 | 3

12. Other Pre Specified Outcome: Number of Participants With Hemodynamic Improvement
Description: Hemodynamic improvement is defined as improvement of ankle-brachial index (ABI) by ≥0.10 or to an ABI ≥0.90 as compared to pre-procedure value without the need for repeat revascularization.
Time Frame: 12 months post procedure
Population: Data for Hemodynamic Improvement are based on subjects with the data point collected.
Measure: Count of Participants; unit: Participants
Arm/Group | DES BTK | Conventional PTA
Number analyzed (Participants) | 91 | 49
Participants | 59 | 28

ADVERSE EVENTS:
Time Frame: Adverse event data collected through 12 months post-index procedure.
Description: All-cause mortality rate is through 12 month visit window (Day 395)
Arm/Group | DES BTK | Conventional PTA
All-Cause Mortality (participants affected / at risk) | 11/130 | 7/71
Serious Adverse Events (participants affected / at risk) | 82/130 | 51/71
Other Adverse Events (participants affected / at risk) | 84/130 | 37/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DES BTK (N=130) | Conventional PTA (N=71)
Peripheral artery stenosis (Vascular disorders) | 12 (24) | 6 (10)
Peripheral artery occlusion (Vascular disorders) | 8 (17) | 5 (6)
Peripheral arterial occlusive disease (Vascular disorders) | 13 (16) | 6 (8)
Peripheral ischaemia (Vascular disorders) | 11 (14) | 5 (7)
Intermittent claudication (Vascular disorders) | 7 (10) | 3 (4)
Peripheral artery thrombosis (Vascular disorders) | 3 (3) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)
Arteriosclerosis (Vascular disorders) | 2 (2) | 0 (0)
Extremity necrosis (Vascular disorders) | 1 (2) | 0 (0)
Embolism arterial (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
May-Thurner syndrome (Vascular disorders) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 10 (11) | 4 (4)
Gangrene (Infections and infestations) | 8 (9) | 1 (1)
Pneumonia (Infections and infestations) | 6 (7) | 2 (3)
Cellulitis (Infections and infestations) | 4 (4) | 2 (3)
Urinary tract infection (Infections and infestations) | 3 (4) | 1 (1)
Localised infection (Infections and infestations) | 3 (3) | 2 (3)
Sepsis (Infections and infestations) | 3 (3) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Abscess limb (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Biliary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Corona virus infection (Infections and infestations) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Diabetic foot infection (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 0 (0)
Scrotal abscess (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Gas gangrene (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 7 (10) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 4 (6) | 0 (0)
Angina pectoris (Cardiac disorders) | 5 (5) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (2) | 2 (2)
Cardiac failure (Cardiac disorders) | 2 (2) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 2 (2) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Vascular procedure complication (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Wound (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Snake bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (5) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ischaemic enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 4 (4) | 2 (4)
Asthenia (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Stent-graft endoleak (General disorders) | 1 (1) | 0 (0)
Ulcer (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic complication (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Marasmus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Shock hypoglycaemic (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 0 (0)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Collagen-vascular disease (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (2) | 1 (1)
Weight decreased (Investigations) | 1 (2) | 0 (0)
Ankle brachial index abnormal (Investigations) | 1 (1) | 0 (0)
Anticoagulation drug level above therapeutic (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Cataract nuclear (Eye disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Toe amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DES BTK (N=130) | Conventional PTA (N=71)
Wound (Injury, poisoning and procedural complications) | 8 (10) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 7 (9) | 1 (4)
Vascular procedure complication (Injury, poisoning and procedural complications) | 4 (5) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Splinter (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 9 (9) | 3 (3)
Peripheral venous disease (Vascular disorders) | 6 (6) | 2 (3)
Intermittent claudication (Vascular disorders) | 3 (6) | 1 (1)
Vasospasm (Vascular disorders) | 4 (5) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 4 (4) | 2 (3)
Hypotension (Vascular disorders) | 3 (3) | 2 (2)
Arterial spasm (Vascular disorders) | 3 (3) | 1 (1)
Reperfusion injury (Vascular disorders) | 3 (3) | 0 (0)
Haematoma (Vascular disorders) | 2 (2) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 4 (4)
Arterial perforation (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 1 (1) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 3 (3)
Cellulitis (Infections and infestations) | 2 (3) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 2 (3) | 1 (1)
Osteomyelitis (Infections and infestations) | 3 (3) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Corona virus infection (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Tinea infection (Infections and infestations) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Wound abscess (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Dermatophytosis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Viral pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 4 (5) | 1 (1)
Chest pain (General disorders) | 3 (3) | 0 (0)
Catheter site bruise (General disorders) | 1 (2) | 0 (0)
Catheter site haematoma (General disorders) | 2 (2) | 0 (0)
Catheter site pain (General disorders) | 2 (2) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 2 (2)
Catheter site related reaction (General disorders) | 1 (1) | 0 (0)
Catheter site swelling (General disorders) | 1 (1) | 0 (0)
Fat necrosis (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Ulcer haemorrhage (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Loose tooth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 (5) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (4)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Plantar erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 2 (3) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Cognitive disorder (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery disease (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Demyelinating Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 2 (2)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Anuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Costovertebral angle tenderness (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Eyelid ptosis (Eye disorders) | 1 (1) | 0 (0)
Scleral disorder (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Inflammatory marker increased (Investigations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Serum ferritin decreased (Investigations) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Device occlusion (Product Issues) | 1 (2) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT03551496/Prot_SAP_000.pdf